CLINICAL TRIAL: NCT07098559
Title: The Effects of Bystander Intervention Model-Based Creative Drama Workshops on Bystander Intervention and Empathy in Peer Bullying Among Middle School Students: A Randomized Controlled Trial
Brief Title: Effects of Bystander Model-Based Creative Drama on Empathy and Bullying Intervention in Middle School Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şeyma Nur HEPOKUR, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-77082166-302.08.01-1265651
Record Dates: First submitted 2025-07-24; First posted 2025-08-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Bystander Intervention
Keywords: creative drama; middle school students; peer bullying; bystander intervention; bystander intervention model; bystander role; emphaty; nursing

STUDY DESIGN:
Intervention Model Description: Randomized study with experimental and control groups
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, it is impossible to blind the researcher implementing the intervention and the participants. A pre-test will be administered before randomization to prevent bias in the study. The study's data collection and statistical process are planned to be blinded. The assignment of students to the intervention and control groups will be made by a statistician independent of the study. The researcher and the students will not know which group they are in until the application begins. After administering the follow-up tests, the independent researcher will code the data as groups A and B and transfer it to SPSS. With this method, the statistician plans to perform analysis and reporting without knowing which group is the intervention group and which is the control group. The codes of the groups are intended to be disclosed after the analysis and reporting of the data. In this way, detection bias, statistical bias, and reporting bias will be prevented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative drama group (Experimental): Participants will be given ten sessions of creative drama intervention training in creative drama workshops reviewed by experts.
  Interventions: Behavioral: Creative drama
- Control group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Behavioral: Creative drama — This intervention is unique in its integration of the Bystander Intervention Model with creative drama techniques to enhance empathy, self-efficacy, and active intervention behaviors among middle school students witnessing peer bullying. Unlike traditional anti-bullying programs that rely on lectures or cognitive-based approaches, this study uses experiential learning and role-playing scenarios to simulate real-life bullying situations and encourage emotional engagement and behavioral change.
  Arms: Creative drama group

SUMMARY:
This research is a randomized controlled experimental study. The research aims to evaluate the effectiveness of creative drama workshops based on the bystander intervention model on middle school students' bystander intervention and empathy levels. The research population consists of sixth and seventh grade students. The research sample will consist of at least 42 middle school students, 21 in the intervention group and 21 in the control group. The sample will be selected through randomization. The students in the intervention group will receive 10 sessions of creative drama intervention. The research aims to answer the following questions: Is there a difference between the intervention group and the control group in terms of bystander intervention levels? Is there a difference between the intervention group and the control group in terms of empathy levels toward the victim of peer bullying?

DETAILED DESCRIPTION:
Adolescence is a crucial period during which individuals undergo significant physical, mental, and social changes, and the process of identity development begins. The transition to middle school during this period leads to increased interaction with peer groups and an increased likelihood of encountering behaviors such as bullying. Bullying, a form of aggression characterized by intent to harm, repetition, and a power imbalance, is a common occurrence in schools. According to a 2023 report by the United Nations Educational, Scientific, and Cultural Organization (UNESCO), one in three students worldwide is bullied, while in Turkey, rates range from 15.9% to 34.9%. Bullying negatively impacts children's physical, mental, and social development, and these effects can extend into adulthood. During bullying, students may assume various roles, including bully, victim, bully-victim, and bystander. Bystander intervention is particularly critical for preventing bullying. However, research shows that a large portion of bystanders remain passive. However, intervening bystanders have the potential to quickly stop bullying. One effective strategy for preventing bullying is school-based, multifaceted intervention programs. The school nurse plays a crucial role in this process, providing guidance both in identifying bullying and in providing intervention. Empathy is a key determinant in bystander intervention. Individuals with high empathy are more likely to take on an advocacy role. In this context, creative drama can increase students' sensitivity to bullying by fostering empathy. Through creative drama, students can experience the effects of bullying and discuss solutions. Drama helps students express their feelings and develop problem-solving and communication skills. The Bystander Intervention Model defines five stages individuals must go through to help a situation: recognizing the incident, interpreting it as urgent, assuming responsibility, knowing how to help, and intervening. Individual attitudes and environmental factors play important roles in this process. In this context, this study aims to evaluate the effectiveness of creative drama workshops based on the bystander intervention model in increasing middle school students' bystander intervention levels and empathy skills in bullying. The study will be conducted with 6th and 7th grade students and will utilize a randomized controlled experimental design. The sample will consist of 42 students, who will be randomly assigned to an intervention group of 21 and a control group of 21. The experimental group will participate in creative drama workshops based on an audience intervention model, while the control group will not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being in 6th or 7th grade,
* Having parental consent, and
* Voluntary participation in the study

Exclusion Criteria:

* Difficulty in reading and writing Turkish, and
* Having a physical/mental disability or illness

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Bystander Intervention Scale in Bullying | 3 months
  The scale aims to evaluate individuals' reactions and attitudes towards bullying incidents they witness and was created based on the Bystander Intervention Model. The scale, consisting of 16 items in total, consists of five sub-dimensions: Noticing the incident, interpreting the incident as a situation requiring immediate help, accepting the responsibility to help, deciding how to intervene, and implementing the intervention decision. The scale, structured as a 5-point Likert-type scale, is applied by rating from "Strongly Disagree" to "Strongly Agree." The overall Cronbach's Alpha reliability coefficient of the scale was calculated as 0.88. The Cronbach's Alpha reliability coefficients for the sub-dimensions are, respectively; 0.60 for recognizing the event, 0.78 for interpreting the event as emergency aid, 0.67 for accepting the responsibility to help, 0.75 for deciding on the intervention method, and 0.78 for implementing the intervention decision

SECONDARY OUTCOMES:
Empathy Scale for Peer Bullying Victims | 3 months
  To assess empathy towards victims of peer bullying. The scale consists of seven items on a five-point Likert-type scale and two subscales: cognitive empathy and affective empathy. The Cronbach's Alpha reliability coefficient for the entire scale is 0.88.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD sharing is restricted by data confidentiality, participant privacy, and applicable ethics rules and legislation. Sharing data with third parties may require relevant ethics committee approval, institutional permissions, and explicit consent from participants. If these conditions are not met, IPD sharing may not be possible.